CLINICAL TRIAL: NCT04087395
Title: A Randomized, Controlled, Double-blinded, Within-subject (Split-face), Multicenter, Prospective Clinical Study to Compare the Level of Pain Using the Dermal Filler RHA® 4 Formulated With Two Different Anesthetics in the Treatment of Nasolabial Folds
Brief Title: RHA® 4 With New Anesthetic - Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TEO-RHA-1802
Record Dates: First submitted 2019-09-02; First posted 2019-09-12 (Actual); Results first posted 2021-06-16 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-05

CONDITIONS: Aging; Pain
Keywords: Hyaluronic Acid; Anesthetic; Lidocaine; Nasolabial Folds
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Split-face design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- RHA®4 with new anesthetic agent (Experimental): Split-face injection of RHA®4 with new anesthetic agent in the nasolabial fold of one side of the face and RHA®4-Lidocaine in the nasolabial fold of opposite side of the face.
  Up to 3 mL injected per side.
  Interventions: Device: RHA®4 with new anesthetic agent
- RHA®4-Lidocaine (Experimental): Split-face injection of RHA®4 with new anesthetic agent in the nasolabial fold of one side of the face and RHA®4-Lidocaine in the nasolabial fold of opposite side of the face.
  Up to 3 mL injected per side.
  Interventions: Device: RHA®4-Lidocaine

INTERVENTIONS:
Device: RHA®4 with new anesthetic agent — A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus zooepidemicus, formulated to a concentration of 23 mg/g and 0.3% w/w of new anesthetic agent in a physiologic buffer.
  Arms: RHA®4 with new anesthetic agent
Device: RHA®4-Lidocaine — A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus zooepidemicus, formulated to a concentration of 23 mg/g and 0.3% w/w lidocaine in a physiologic buffer.
  Arms: RHA®4-Lidocaine

SUMMARY:
This is a randomized, controlled, double-blinded, within-subject (split-face), multicenter, prospective study to investigate whether RHA® 4 with New Anesthetic Agent is non-inferior to RHA® 4 (with lidocaine) in terms of injection site pain felt by the subject during injection.

At screening, the Treating Investigator (TI) evaluated subjects' NLF severity (using the Wrinkle Severity Rating Scale; WSRS) to confirm eligibility and to establish a pre-treatment score for assessing aesthetic improvement.

At Visit 1, RHA® 4 With New Anesthetic Agent was administered in a random sequence (first or second injection) and side of the face (left or right) and RHA® 4 with lidocaine was administered to the other side. Study subjects and the TI injecting study devices were blinded.

Immediately after injection of each side, subjects rated injection site pain experienced during injection using a 100 mm Visual Analog Scale (VAS). Injection site pain in each side of the face was also assessed at 15, 30, 45 and 60 minutes post-injection.

Safety evaluation consisted of AE assessments, a 30-day CTR (Common Treatment Response) diary and a follow-up call performed by the study site at 72 hours after injection.

Subjects attended Visit 2 (30 days post-injection) where efficacy and safety assessments will be conducted. Subjects who present with an unresolved clinically significant device related AE at Visit 2 received the optional follow-up phone call no later than 30 days after Visit 2. If the clinically significant AE remained unresolved, the Investigator requested that the subject attended the optional in-clinic follow-up visit (i.e., Visit 3) within 5 working days. Follow-up of the clinically significant AE continued until the AE was resolved or the TI determines that additional follow-up was not necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient, male or female of any race, 22 years of age or older. Female subjects of childbearing potential must have a negative UPT at Visit 1 and practice a reliable method of contraception throughout the study.
2. Moderate to severe bilateral nasolabial folds (grade 3 or 4 on the five-point WSRS).
3. Nasolabial folds of the same WSRS grade on the left and right sides of the face.
4. Able to follow study instructions and complete all required visits.
5. Sign the IRB-approved ICF, Photographic Release Form, the Authorization for Use and release of Health and Research Study Information (HIPAA) form, and if applicable the California Experimental Research Subject's Bill of Rights prior to any study-related procedures being performed.

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding, or of childbearing potential and not practicing reliable birth control.
2. Known hypersensitivity or previous allergic reaction to any component of the study devices.
3. Use of a prohibited treatment/procedure within time periods defined in the protocol
4. Known sensitivity to local anesthetics of the amide type, history of multiple severe allergies, or history of anaphylactic shock.
5. History of active chronic debilitating systemic disease that, in the opinion of the investigator, would make the subject a poor candidate in the study.
6. History of connective tissue disease.
7. Malignancy (excluding non-melanoma skin cancer) within the past 5 years.
8. History of skin cancer in the treatment area.
9. Clinically active disease or infection in the NLF area.
10. Medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with the interpretation of study results or compliance of the subject and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.
11. Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.
12. Exposure to any other investigational drug/device within 90 days of entering the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - California, Beverly Hills, California
  - Florida, Coral Gables, Florida
  - Illinois, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Groups:
- Split-face Study : Bilateral Treatment RHA® 4 With New Anesthetic Agent Vs RHA® 4-Lidocaine: Split-face injection of RHA® 4 with new anesthetic agent in the NLF on one side of the face and RHA® 4- Lidocaine in the NLF on the opposite side of the face.
  RHA® 4 with new anesthetic agent was administered in a random sequence (first or second injection) on one side and RHA®4-Lidocaine was administered in the side.
Period: Overall Study
Arm/Group | Split-face Study : Bilateral Treatment RHA® 4 With New Anesthetic Agent Vs RHA® 4-Lidocaine
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Split-face Study : Bilateral Treatment With RHA®4 With New Anesthetic Agent Vs RHA®4-Lidocaine: Split-face injection of RHA®4 with new anesthetic agent in the nasolabial folds on one side of the face and RHA®4-Lidocaine in the perioral rhytids on the opposite side of the face
Arm/Group | Split-face Study : Bilateral Treatment With RHA®4 With New Anesthetic Agent Vs RHA®4-Lidocaine
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick scale is a numerical classification schema for human skin color:
  Type I - always burns, never tans (pale white; blond or red hair; blue eyes; freckles); Type II - usually burns, tans minimally (white; fair; blond or red hair; blue, green, or hazel eyes); Type III - sometimes mild burn, tans uniformly (cream white; fair with any hair or eye color); Type IV - burns minimally, always tans well (moderate brown); Type V - very rarely burns, tans very easily (dark brown); Type VI - Never burns, never tans (deeply pigmented dark brown to darkest brown)
  Participants
    Types I to III (as assessed by TI at screening) | 19
    Types IV to VI (as assessed by TI at screening) | 11

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority of RHA® 4 With New Anesthetic Agent Versus RHA® 4-Lidocaine in Terms of Reducing Pain During Device Injection Into Nasolabial Folds.
Description: Injection pain during injection will be based on the 100 mm Visual Analog Scale (VAS), as assessed by subjects immediately after injection of each nasolabial fold.
  VAS is a 100 mm Visual Analog Scale with 0 meaning no pain and 100 meaning intolerable pain.
Time Frame: Visit 1 - During Injection
Measure: Mean (Standard Deviation); unit: mm
Groups:
- RHA®4 With New Anesthetic Agent; RHA®4-Lidocaine: Split-face injection of RHA®4 with new anesthetic agent in the nasolabial fold of one side of the face and RHA®4-Lidocaine in the nasolabial fold of opposite side of the face.
Arm/Group | RHA®4 With New Anesthetic Agent | RHA®4-Lidocaine
Number analyzed (Participants) | 30 | 30
mm | 17.1 (18.38) | 16.3 (18.89)
Statistical Analysis 1: Comparison: RHA®4 With New Anesthetic Agent vs RHA®4-Lidocaine; Test type: Non-Inferiority — To achieve non-inferiority, the observed p-value must be <= 0.5 taking into account of the non-inferiority margin (i.e., 10mm difference in Pain VAS between the two treatment groups); p < 0.0001, t-test, 1 sided — One-sided paired student t-test

2. Secondary Outcome: Difference Between RHA® 4 With New Anesthetic Agent Versus RHA® 4-Lidocaine in Term of Reducing Pain at 15, 30, 45 and 60 Minutes Post-injection in Nasolabial Folds of Each Side of the Face.
Description: Injection pain was measured on the 100 mm Visual Analog Scale (VAS), as assessed by subjects in nasolabial fold of each side of the face.
  VAS is a 100 mm Visual Analog Scale with 0 meaning no pain and 100 meaning intolerable pain
Time Frame: Visit 1 - 15, 30, 45 and 60 minutes post-injection
Measure: Mean (Standard Deviation); unit: mm
Groups:
- RHA®4 With New Anesthetic Agent: Split-face injection of RHA®4 with new anesthetic agent in the nasolabial fold of one side of the face and RHA®4-Lidocaine in the nasolabial fold of opposite side of the face.
  Up to 3 mL injected per side.
  RHA®4 with new anesthetic agent: A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus zooepidemicus, formulated to a concentration of 23 mg/g and 0.3% w/w of new anesthetic agent in a physiologic buffer.
- RHA®4-Lidocaine: Split-face injection of RHA®4 with new anesthetic agent in the nasolabial fold of one side of the face and RHA®4-Lidocaine in the nasolabial fold of opposite side of the face.
  Up to 3 mL injected per side.
  RHA®4-Lidocaine: A sterile, biodegradable, biocompatible, viscoelastic, clear, colorless, homogenized gel implant. It consists of cross-linked hyaluronic acid produced by fermentation of Streptococcus zooepidemicus, formulated to a concentration of 23 mg/g and 0.3% w/w lidocaine in a physiologic buffer.
Arm/Group | RHA®4 With New Anesthetic Agent | RHA®4-Lidocaine
Number analyzed (Participants) | 30 | 30
mm
  15 Min | 4.9 (12.33) | 5.1 (15.94)
  30 Min | 2.0 (5.66) | 3.1 (12.30)
  45 Min | 0.0 (0.00) | 2.1 (11.68)
  60 Min | 0.0 (0.00) | 1.9 (10.22)

3. Secondary Outcome: Change in NLF WSRS Score Between Baseline and Day 30 as Assessed by the Treating Investigator
Description: NLF-WSRS (Nasolabial Folds- Wrinkle Severity Rating Scale) is a validated 5-grade scale with 1 being "Absent" and 5 being "Extreme"
Time Frame: Visit 1 - Baseline (pre-injection), Visit 1 (post-injection), Visit 2 (Day 30)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RHA®4 With New Anesthetic Agent | RHA®4-Lidocaine
Number analyzed (Participants) | 30 | 30
units on a scale
  Visit 1 (post-injection) | -1.8 (0.57) | -1.8 (0.57)
  Visit 2 (Day 30) | -1.9 (0.48) | -1.8 (0.63)

4. Secondary Outcome: Percentage of Responders Based on the Intra-individual Improvement of at Least One Grade on the Nasolabial Folds Wrinkle Severity Rating Scale (NLF-WSRS) Compared to Baseline, as Assessed by the TI
Description: A responder corresponds to a subject with an intra-individual improvement of at least one grade on the NLF WSRS compared to Baseline, as assessed by the TI
Time Frame: Visit 1 (Baseline, pre-injection), Visit 1 (post-injection), Visit 2 (Day 30)
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 With New Anesthetic Agent | RHA®4-Lidocaine
Number analyzed (Participants) | 30 | 30
Participants
  Visit 1 (post-injection): Responder | 30 | 30
  Visit 1 (post-injection): Not Responder | 0 | 0
  Visit 2 (Day 30): Responder | 30 | 29
  Visit 2 (Day 30): Not Responder | 0 | 1

5. Secondary Outcome: Subject's Perception of Treatment Effectiveness as Per the FACE-Q (Nasolabial Folds Domain) Questionnaire. The FACE-Q Measures the Experience and Outcomes of Aesthetic Facial Procedures From the Patient's Perspective.
Description: FACE-Q questionnaire is composed of 5 questions with a score linked to answers (1 being 'Not at all' and 4 being 'Extremely').
  The subject will be instructed as follows: "These questions ask about how you look right now. For each question, circle only one answer. With your nasolabial folds in mind (the deep lines that run downward from the sides of your nose), in the past week, how much have you been bothered by:", and will provide response.
  To calculate the FACE-Q, outcomes from all 5 questions were pooled, data were transformed so that higher scores reflected a superior outcome, and adapted to a scale of 100 units (i.e. lowest score = 0, highest score = 100).
Time Frame: Visit 1 (Baseline) and Visit 2 (Day 30)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHA®4 With New Anesthetic Agent | RHA®4-Lidocaine
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline Face-Q Score | 25.2 (21.12) | 24.3 (20.34)
  Day 30 Face-Q Score | 89.0 (15.19) | 88.5 (16.16)
  Face-Q Change from Baseline to Day 30 | 63.8 (24.69) | 64.2 (25.06)

6. Secondary Outcome: Number of Subjects Scored Either "Much Improved" or "Improved" on Global Aesthetic Improvement (GAI) by the Treating Investigator (TI)
Description: Global Aesthetic Improvement (GAI) is a subjective 5-grade scale comprised of "much improved, improved, no change, worse, and much worse".
  GAI was assessed using the baseline photograph. Each side of the face will be assessed independently.
Time Frame: Visit 1 (just after receiving treatment) and Visit 2 (Day 30)
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 With New Anesthetic Agent | RHA®4-Lidocaine
Number analyzed (Participants) | 30 | 30
Participants
  Visit 1 (post-injection) | 30 | 30
  Visit 2 (Day 30) | 30 | 29

7. Secondary Outcome: Number of Global Aesthetic Improvement (GAI) Responders (i.e., Scoring Either "Much Improved" or "Improved") on GAI Scale According to Subject's Self-assessment
Description: Global Aesthetic Improvement (GAI) is a subjective 5-grade scale comprised of "much improved, improved, no change, worse, and much worse".
  GAI was assessed using the baseline photograph. Subjects were instructed: "Use a mirror to compare your face to the photograph provided to you and rate the degree of aesthetic improvement by using the following scale".
  Each side of the face was assessed independently.
Time Frame: Visit 1 (just after receiving treatment) and Visit 2 (Day 30)
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 With New Anesthetic Agent | RHA®4-Lidocaine
Number analyzed (Participants) | 30 | 30
Participants
  Visit 1 (post-injection) | 30 | 30
  Visit 2 (Day 30) | 30 | 30

8. Secondary Outcome: Number of Subjects "Satisfied" or "Very Satisfied" With Study Treatment Using the Subject's Satisfaction Scale
Description: The Subject Satisfaction Scale is a subjective, balanced, 5-point scale assessing subject satisfaction with study treatment. Possible scores range from with 1 (very satisfied) to 5 (very dissatisfied).
  Proportion of subjects who were Satisfied (i.e., 1-Very Satisfied + 2-Satisfied) was compared to the proportion of subjects who were Not Satisfied (i.e., 3-Neither Satisfied nor dissatisfied + 4-Dissatisfied + 5-Very Dissatisfied)
Time Frame: Visit 1 (just after receiving treatment) and Visit 2 (Day 30)
Measure: Number; unit: participants
Arm/Group | RHA®4 With New Anesthetic Agent | RHA®4-Lidocaine
Number analyzed (Participants) | 30 | 30
participants
  Visit 1 (post-injection) : Satisfied | 30 | 30
  Visit 1 (post-inj): Not Satisfied | 0 | 0
  Visit 2 (Day 30) : Satisfied (i.e., 1-Very Satisfied + 2-Satisfied) | 29 | 29
  Visit 2 (Day 30) : Not Satisfied | 1 | 1

9. Secondary Outcome: Number of Subjects With Post Injection Treatment Responses (From Common Treatment Responses (CTR) Diary) for Safety Evaluation of RHA® 4 With New Anesthetic Agent Versus RHA® 4-Lidocaine
Description: The subjects received a diary booklet and instructions for recording their observations of the Common Treatment Responses to the study treatments during 30 days following the injection. The diary were discussed during follow-up phone call and visit. Subjects were instructed to complete the diary at approximately the same time each day (i.e., am or pm).
  The subject diary captured the following Common Treatment Responses (CTR) that occur following the injection of a dermal filler; specifically, redness, pain, tenderness, firmness, swelling, lumps/bumps, bruising, itching, discoloration, and "other".
  The 30-day patient CTR diary included a detailed glossary describing all signs/symptoms listed in the diary; an option was provided to rate "other" if the subject experienced a sign/symptom that is not listed.
Time Frame: During 30 days after injection
Measure: Count of Participants; unit: Participants
Arm/Group | RHA®4 With New Anesthetic Agent | RHA®4-Lidocaine
Number analyzed (Participants) | 30 | 30
Participants
  Bruising | 19 | 21
  Discoloration | 11 | 12
  Firmness | 24 | 22
  Itching | 7 | 6
  Lumps/Bumps | 22 | 21
  Pain | 12 | 9
  Redness | 21 | 20
  Swelling | 21 | 23
  Tenderness | 24 | 24
  Paresthesia | 1 | 0

ADVERSE EVENTS:
Time Frame: approximatly 1 month (35 days, overall study duration)
Arm/Group | RHA®4 With New Anesthetic Agent | RHA®4-Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 4/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RHA®4 With New Anesthetic Agent (N=30) | RHA®4-Lidocaine (N=30)
Injection site induration (General disorders) | 3 (3) | 4 (4)
Injection site mass (General disorders) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 1 (1)
Paresthesia oral (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT04087395/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT04087395/SAP_001.pdf